# 临床研究方案

项目名称: 髌腱联合筋膜手法协调中心点的体外冲击波治疗髌腱

炎的临床疗效:一项随机对照试验

申请单位:中山大学孙逸仙纪念医院

版本号: V2.0

版本日期: 2025.12.21

项目负责人: 柯松坚

方案签字确认: 极 办 湿.

### 合规性声明

遵守《药物临床试验质量管理规范》 以及 《医疗卫生机构开展研究者发起的临床研究管理 办法》的规定及赫尔辛基宣言,承诺依照此方案实施本研究,参与者必须经过培训,在获得伦理 委员会书面批准及受试者书面知情同意后实施研究,方案修订需重新通过批准。

注:本模板为干预性研究模板,其他研究类型请根据项目实际需求对符号"\*"标注的内容进行修改或删减。

一、方案摘要(题目、研究简要描述、研究对象、结局指标、研究干预\*、样本量等,字数在 300-500 字)

髌腱炎(patellar tendonitis,pt),又称跳跃膝,主要表现为髌前酸胀、疼痛,严重者影响患者的生活质量。临床上髌腱炎以保守治疗为主,而体外冲击波疗法(ESWT),通过对髌腱进行痛点处理,可有效缓解与软组织相关的疼痛和松解软组织粘连;许多研究已证实其短期疗效,但其中期维持效果尚未明确。意大利筋膜手法(fascial manipulation,FM)基于身体一体化理论,从筋膜相互影响的原则,采用结构化的评估以识别髌腱周围特定筋膜致密化区域,通过消除筋膜致密化,恢复筋膜组织生理张力并促进层间正常滑动,减轻髌腱炎患者患膝负荷、防止疼痛加重。体外冲击波治疗(ESWT)通过高频振动,具有松解筋膜的作用,可同样影响筋膜链,因此本研究拟纳入38名诊断为髌腱炎且满足体外冲击波治疗适应症的患者,在入组和获得知情同意后采用随机数字表进行随机分为试验和对照组,根据分组情况分别给予髌腱联合筋膜手法协调中心点冲击波治疗及单纯髌腱冲击波治疗。在基线、所有治疗完成后当天、所有治疗结束后第1个月、第3个月收集数据,进行统计分析,比较治疗前后的数据变化值差异,评估髌腱联合筋膜手法协调中心点的体外冲击波治疗髌腱炎的短期和中期维持疗效是否优于单纯髌腱体外冲击波治疗组,为髌腱炎治疗提供更优化的治疗方案。

### 二、引言(引言资料中应标注引用的参考文献)

2.1 研究理论基础/背景(从疾病、治疗标准和已知治疗的局限阐述为什么要进行临床研究,以及说明临床前研究、药理学研究和相关研究的发现、研究的重要性)

髌腱炎是指连接髌骨与胫骨的髌腱因反复过度负荷导致的无菌性炎症或退行性病变,也被称为髌腱病(patellar tendinopathy),常见髌骨下极(髌腱近端)疼痛,严重时可牵涉至髌下区域;同时可伴随肿胀、膝关节无力等症状。组织病理学显示,髌腱由于长期承受重复牵拉应力(如跳跃、急停动作),导致胶原纤维出现微撕裂,逐渐积累,最终髌腱发生黄褐色变性和钙化。因此,多数证据强调髌腱炎的本质是退行性肌腱病(tendinopathy),而非急性炎症。髌腱炎患者步行过程中倾向于减少膝、踝屈曲以规避疼痛,但反而增加地面反作用力

(GRF)和关节力矩,形成恶性循环。同时,即使单侧发病,健侧也可能出现生物力学代偿(如步态不对称),增加双侧损伤风险。为分担疼痛处的负荷,股四头肌肌腱及髂胫束可能代偿性增厚,但过度代偿反而加重髌腱应力,髌腱也出现弹性模量降低,从而导致全身性筋膜适应性改变。筋膜链的张力失衡,又进一步影响髌腱负荷[1-2]。

临床上髌腱炎的保守治疗手段包括服用抗炎药、局部注射、支具固定、运动疗法、手法治疗、肌内贴扎技术、体外冲击波疗法 (ESWT)、激光和超声波治疗等,但目前证据显示口服非甾体药物的治疗效果维持较短,而离子电渗疗法、按摩、电疗、运动锻炼和皮质类固醇注射等治疗容易复发[3-4]。这些治疗手段中大部分都是针对髌腱区域组织进行消炎止痛的,只有体外冲击波针对髌腱去进行刺激性治疗,刺激肌腱的修复和组织再生。

近年来,体外冲击波疗法(ESWT)以其修复作用在治疗髌腱炎等肌腱病中的应用激增。冲击波疗法被认为可以通过新生血管形成、细胞增殖和抗炎作用等多种机制刺激慢性肌腱病的组织修复和再生,并减轻局部的疼痛和降低敏感性。大部分研究通过对髌腱周围痛点进行治疗,可有效缓解疼痛和提高膝关节功能,是治疗髌腱炎的有效手段,但部分中期维持疗效尚未明确[5-14]。

意大利筋膜手法(fascial manipulation, FM)基于身体一体化理论,从筋膜相互影响的原则,采用结构化的评估以识别髌腱周围特定筋膜致密化区域,消除筋膜致密化,恢复筋膜组织生理张力并促进层间正常滑动,在减轻髌腱炎患者患膝负荷、改善患侧下肢生物力学、防止疼痛加重方面体现出非常大的潜力<sup>[15-16]</sup>。 因此,筋膜手法也被证实可缓解髌腱炎疼痛。

体外冲击波治疗(ESWT)治疗原理是导子通过对靶区的高速震动进行松解筋膜,可同样改善筋膜链的异常张力。因此本研究探讨基于筋膜理论,采用髌腱联合筋膜手法协调中心点进行体外冲击波治疗,观察其治疗效果是否优于单纯髌腱痛点治疗方案,通过改变筋膜异常张力以维持更长时间的治疗效果。

- 2.2 风险/获益评价
- 2.2.1 已知潜在风险

冲击波治疗的风险:

(1) 冲击波治疗相关并发症:包括治疗后24小时内局部软组织肿胀、瘀血、

皮肤破损、痛性晕厥等。

- (2) 过度炎症反应: 冲击波治疗后短期内可能诱发一过性炎症反应,导致治疗后 24 小时至 48 小时内疼痛加重。
- (3)治疗效果不一: 髌腱炎患者因年龄、病因、病程等个体化原因导致冲击波治疗效果可能出现不一致。

### 2.2.2 已知潜在效益

冲击波治疗的获益:

- (1)减轻疼痛:冲击波能量可以抑制疼痛感受器的敏感性,减少 P 物质,促进 NO 释放,从而缓解髌腱处疼痛。
- (2)促进组织修复与微循环:冲击波通过压力波作用于髌腱,在组织界面产生拉应力和压应力,松解粘连组织,促进局部血管新生,改善血液循环,加速炎症消退和组织修复。此外,冲击波能刺激细胞氧摄入,促进胶原蛋白合成,增强肌腱弹性。
- (3) 松解筋膜:冲击波在筋膜处产生拉应力和压应力,使局部筋膜组织产生弹性变形,改善深部肌肉筋膜的致密化,恢复整体筋膜链的张力平衡。
- (4) 促进筋膜组织的再生:通过刺激成纤维细胞的活性,加速筋膜胶原蛋白的重组和再生,促进正常的筋膜组织恢复。
- (5) 改善下肢运动功能:通过对筋膜的处理则能起到手法类似的作用,改善引起髌腱区域损伤后筋膜不正常的张力,恢复整个下肢筋膜链正常的生物力学,改善下肢的运动表现。
- (6)减少镇痛药物依赖:可能更快更持久地解决患者疼痛的困扰,减少对镇痛药物(如 NSAIDs)的依赖,从而减少药物副作用。

### 2.2.3 潜在风险效益评价

冲击波治疗的潜在风险效益评价:

- (1) 潜在风险: 冲击波治疗过程中可能会导致患者出现熟悉的疼痛而不被接受导致治疗中断;
- (2)潜在效益:探索髌腱联合筋膜手法协调中心点的冲击波治疗对髌腱炎患者的疗效,可能找到一种更有效的冲击波治疗髌腱炎的方法。
  - (3) 潜在风险效益评价:治疗前充分告知治疗过程中和治疗后可能出现的

不适,签署知情同意书,进行髌腱联合筋膜手法协调中心点的冲击波治疗。相比 于小小的风险,后续获得的治疗效益、经济效益和社会效益可能更高,值得进行 探索。

三、研究目的和终点(列表阐述目的(要解决的具体问题),与结局指标对应)

### 3.1目的

#### 3.1.1 主要目的

评估髌腱联合筋膜手法协调中心点体外冲击波治疗髌腱炎在缓解疼痛方面 的有效性和持久性,明确在髌腱炎的冲击波治疗中联合协调中心点的治疗思路是 否优于传统的痛点(单纯髌腱)治疗。

### 3.1.2 次要目的

探究联合筋膜手法协调中心点体外冲击波治疗,对比传统治疗思路体外冲击 波治疗髌腱炎过程中缓解疼痛的短期疗效、对髌腱厚度的影响以及改善膝关节功能障碍的治疗效果。

### 3.1.3 探索性目的

探究髌腱炎冲击波治疗中的一种更加持久高效的方法。

### 3.2 研究指标

### 3.2.1 主要指标及定义

治疗前后的疼痛缓解程度的中期维持效果。使用视觉模拟评分(VAS)来定量评估治疗后随访3个月的疼痛强度变化值。在基线和所有治疗完成后第3个月,由经过培训的不参与干预治疗及数据分析的治疗师使用视觉模拟评分量表评估。

### 3.2.2 次要指标及定义

- (1) 患者膝关节髌腱厚度的变化值:在基线、所有治疗完成后当天,由经过培训的不参与干预治疗及数据分析的治疗师使用便携式肌骨超声成像系统进行患者患侧膝关节髌腱厚度的评估。
- (2) 患者膝关节功能的变化值:在基线、所有治疗完成后当天、所有治疗完成后第1个月及第3个月,由经过培训的不参与干预治疗及数据分析的治疗师使用 Lysholm 膝关节评分量表进行患者患侧膝关节功能的评估。

(3) 患者膝关节疼痛强度的早期变化值:在基线、所有治疗完成后当天和所有治疗完成后第1个月,由经过培训的不参与干预治疗及数据分析的治疗师使用视觉模拟评分量表评估。

### 3.2.3 安全性指标

包括治疗途中或治疗后出现严重皮损、局部严重肿胀、严重痛性晕厥等严重不良事件。

### 四、研究人群

#### 4.1 入选标准

- (1) 年龄为 18 至 45 岁的成年人:
- (2)符合《实用运动医学》(2023版)髌腱炎诊断标准;
- (3) 膝关节疼痛 VAS 评分≥3 分及≤7 分;
- (4) 无其他影响下肢力量或行走的骨科或神经系统疾病:
- (5) 自愿签署知情同意书,并能够配合本研究的治疗和随访。

### 4.2 排除标准

- (1) 一年内膝关节手术史;
- (2) 存在其他原因导致的膝关节前侧疼痛,或有累及膝关节疼痛性疾病或影响 关节的疾病(包括但不限于:一过性滑膜炎、骨结核、骨肿瘤、急性创伤性关节 炎、化脓性关节炎、类风湿性关节炎、代谢性骨病、银屑性关节炎、痛风性关节 炎、骨坏死、强直性脊柱炎或活动性感染等):
- (3) 存在因其他原因引起的膝关节的慢性疼痛(如带状疱疹后神经痛、骨质疏松等);
- (4)使用冲击波治疗的禁忌症,例如:下肢深静脉血栓、出血性疾病或凝血功能障碍、妊娠、认知功能障碍等;
- (5) 有癌性肿瘤、严重支气管扩张、急性化脓性炎症、高烧、活动性肺结核、 心力衰竭、严重贫血、脑血管疾病,或体内植入心脏起搏器等;
- (6)由于其他健康问题无法参与试验,如突发严重外伤、突发严重传染性疾病等。
- 4.3 生活方式注意事项(生活方式有关的限制条件:吸烟、饮酒、运动、饮食等方面,以及如果受试者需要使用方案中禁止使用的药物、治疗或手术时,将采取

### 何种处理措施)

患者入组后出现如下情况将无法继续参加试验: 1. 使用关节内或口服皮质类 固醇药物; 2. 突发原因需行膝关节或髋关节手术; 3. 患者自我体育锻炼时间发生 明显变化。

4.4 筛选失败(对于筛选失败的定义、以及如何处理筛选失败研究对象) 无

4.5 招募和保留策略(如何招募受试者(地点、方式、预期人数.....);如何保留受试者(多种联系方式、激励);如涉及弱势群体:理由+保障措施;如有补偿或激励措施:对象、数量、形式、时间等)

科室门诊或住院髌腱炎患者,经入选标准和排除标准筛选后,详细告知研究 方案、风险,及签署知情同意书。

本研究中,冲击波治疗为非免费治疗项目,患者评估和健康教育为免费项目。 同时,所有入组患者有专人联系通知随访和治疗时间,专门治疗师负责评估和对 患者进行健康教育。

### 五、研究设计

- 5.1 总体设计(包括假设、类型等) 前瞻性、随机双盲对照。
- 5.2 研究设计流程
- 5.2.1 研究具体实行流程

本研究为随机对照试验。纳入诊断为髌腱炎且满足冲击波治疗适应症的患者。在入组和获得知情同意后进行相关临床资料和评估的采集。采用随机数字表进行随机分组:试验和对照组。根据分组情况,试验组给予髌腱联合筋膜手法协调中心点体外冲击波治疗,对照组仅给予单纯髌腱体外冲击波治疗。治疗由一名有丰富临床经验的康复科治疗师完成。在基线、所有治疗完成后当天使用 Visual Analogue Scale (VAS) 评分、Lysholm 膝关节评分量表进行受试者疼痛和膝关节功能等数据的采集,使用便携式肌骨超声成像系统进行患者患侧膝关节髌腱厚度的数据采集;在所有治疗结束后第1个月、第3个月使用 Visual Analogue Scale (VAS) 评分、Lysholm 膝关节评分量表进行受试者的疼痛和膝关节功能的

随访评估并采集数据。

- 5. 2. 2 研究流程图 1
- 5.2.3 研究日程表 2
- 5.3 减少偏倚的方法(例如:随机化、盲法、匹配方法等)

本研究采用计算机软件随机生成数字,将符合入选标准的受试者以 1:1 比例分配到两组。随机码装入不透明、封闭的信封,由专职统计员在受试者进入试验后现场抽取,这样受试者在进入治疗前就无法得知自己属于哪一组。

使用同一型号的体外冲击波仪,设定相同的能量、频率和治疗时长。仪器在两组均产生相同的噪声和振动感,使受试者仅凭感觉难以辨别治疗部位。为避免受试者通过视觉辨认部位,治疗时在膝关节及大腿前侧均覆盖不透光的无菌敷料或遮蔽帘,仅露出探头接触的皮肤区域。这样每位受试者在整个疗程中接受的"感受"基本相同,难以判断自己属于哪一组。

选用外观相同、内部填充吸能材料,能够保持同样的噪声与振动的安慰剂探头。治疗分为三段进行,每位受试者先接受髌腱处 2000 次治疗,接着接受髌腱处 4000 次治疗,最后接受筋膜手法协调中心点 4000 次治疗,每段治疗中间休息 1 分钟。每次休息期间,受试者和负责治疗的物理治疗师离开治疗房间后,由专门的技术员进入房间根据随机分组抽取的随机码情况进行决定是否更换安慰剂探头。装配探头后技术员立即离开房间,过程中避免与患者和负责治疗的物理治疗师碰面导致暗示。之后受试者和负责治疗的物理治疗师继续进入房间进行治疗。全程技术员和受试者以及负责治疗的物理治疗师均不知道受试者所属组别。

受试者的评估和随访由独立的物理治疗师完成,他们在整个试验期间对受试者的分组信息保持盲态,评估工具(如 VAS、Lysholm 膝关节评分量表、超声检查等)均在统一的环境下进行。

在每次随访结束后,要求受试者和评估者分别猜测自己所属的组别,并记录 猜测正确率。

所有原始数据使用编码方式保存,统计分析由未接触分组信息、不清楚受试者分组情况的负责统计的统计师完成。分析报告在解盲前仅提供总体均值、方差等汇总信息。

通过以上方法去减少该试验的偏倚。

- 5.4 研究结束的定义(例如:最后一个研究对象完成最后一次随访)研究结束的定义为:最后一个研究对象完成最后一次随访。
- 5.5 统计分析

### 5.5.1 样本量及计算依据

查阅文献数据<sup>[17]</sup>,参考文献中干预治疗后 3 个月时,试验组和对照组患者 VAS 评分相对于基线的变化值的预期均值差  $\Delta$  =2. 0,标准差(SD)  $\sigma$  为 2. 5。

考虑到基线值对终点结局有显著影响,采用 ANCOVA,将基线 VAS 评分作为协变量进行调整后,残差标准差通常会降低。降低的幅度与基线值和终点值的相关系数( $\rho$ )有关,即 $\sigma_{\text{ANCOVA}} = \sigma \cdot \sqrt{1-\rho^2}$ 。根据参考文献研究,调整后的残差标准差为原始 SD 的 80%,即 $\sigma_{\text{ANCOVA}} = 2.5 \cdot 0.8 = 2.0$ 。

根据本临床试验研究 1 : 1(试验组 : 对照组)的设计,结合主要疗效结局指标,基于 ANCOVA 的优化估算,假设本研究的 I 类错误概率  $\alpha=0.05$ ,把握度  $(1-\beta)=80\%$ ,采用如下公式进行样本量估算: $n_{per-group}=\frac{2\cdot \left(Z_{\partial/2}+Z_{\beta}\right)^2\cdot \sigma^2}{\Delta^2}$ ,估算本研究所需要的样本量,两组共需招募 32 名受试者,每组 16 人。

考虑试验过程中 15%的脱落率,采用如下公式进行调整:  $n_{adjusted-per-group} = \frac{n_{per-group}}{1-D}$ ,最终确定总样本量为 38 人 。

### 5.5.2 数据分析集(如全分析集、符合方案集、安全性分析集)

本研究采用意向性治疗原则进行分析。所有经过随机化的患者(全分析集,FAS)均被纳入主要疗效分析。同时,我们也定义了符合方案集(PPS),该集合排除了存在重大方案违背的患者,用于支持性分析。安全性分析在所有至少接受过一次研究冲击波治疗的患者(安全性分析集,SS)中进行。主要疗效指标(治疗后3个月VAS评分变化值)的缺失数据采用**多重填补法**进行处理。

### 5.5.3 统计分析计划

统计分析的资料描述、主要指标/次要指标/安全性指标的分析方法、统计学校正方法、偏倚的控制、分层/亚组/敏感性分析等

本研究会明确缺失值的可能来源(随访失访、测量错误等),并预设缺失机制(MCAR、MAR),采用 MICE 进行多重插补进行缺失数据的处理。对于连续的功能评分(如 VAS)使用线性回归插补;对分类变量(如治疗组别、性别)使用

逻辑回归或多项式回归。设置 m=5 次插补,以平衡计算负担与估计精度。

本研究采用 SPSS 27.0 对数据进行整理和统计学分析。在此过程中,我们以 P<0.05 作为差异有统计学意义的标准。对年龄、治疗前后的 VAS 评分及 Lysholm 膝关节评分、治疗前后的髌腱厚度等计量资料进行探索性分析判断其是 否符合正态分布。若符合正态分布,则采用均数土标准差进行统计描述;若不符合正态分布,则采用中位数和四分位数间距进行描述。性别计数资料采用频数进行描述。

本研究采用差异性检验,计量资料(VAS,Lysholm 膝关节评分、髌腱厚度)采用均数±标准差,计数资料(性别,不良事件报告数)采用百分率。最后一次的缺失值用以前的值来代替,计量资料(VAS,Lysholm 膝关节评分、髌腱厚度)的组间比较用 t 检验(若服从正态分布),而计数资料(性别,不良事件报告数)的组间比较用卡方检验或 Fisher 精确概率检验(视具体情况);。观察比较两组样本的治疗前后的指标差异以及组间差异。P < 0.05 认为有统计学意义。

治疗前基线数据比较:

治疗前两组间的 VAS 评分、Lysholm 膝关节评分、患侧膝关节髌腱厚度,通过探索性分析判断其是否符合正态分布。若符合正态分布,采用独立样本 t 检验进行统计比较;若不符合正态分布,则采用 Mann-Whitney U 秩和检验进行统计比较。性别采用卡方检验比较两组分类变量的均衡性。

干预后组间比较方法:

两组间的 VAS 评分变化值、Lysholm 膝关节评分变化值、患侧膝关节髌腱厚度变化值,通过探索性分析判断其是否符合正态分布。若符合正态分布,采用独立样本 t 检验进行统计比较;若不符合正态分布,则采用 Mann-Whitney U 秩和检验进行统计比较。

组内比较方法(干预前后):

符合正态分布的数据: 配对 t 检验

非正态分布数据: Wilcoxon 符号秩检验

对干预前后两组内研究对象的 VAS 评分、Lysholm 膝关节评分、患侧膝关节髌腱厚度计量资料及各指标治疗前后的差值进行正态性检验,治疗前后及差值均符合正态分布的指标,则采用配对样本 t 检验进行统计对比;若不符合正态

分布,则采用 WilcoxonSigned-RankTest 进行统计对比。

本研究的安全性评价主要围绕不良事件(AE)展开,分析方法以描述性统计为主,具体步骤如下:

确定安全性指标(不良事件):记录每例患者在治疗期间出现的任何不良反应,包括局部疼痛、皮肤红肿、痛性眩晕等:

数据收集与整理:在每次冲击波治疗期间记录患者自述的不良反应,建立病例报告表,每行对应一例患者,列包括:患者编号、性别、年龄、病程、治疗方案、每次 AE 出现时间、AE 类型、AE 等级等。

描述性统计指标(不良事件发生率):发生率= $\frac{\text{出现AE} \, \text{的患者数}}{\text{总患者数}} \times 100\%$ ,依据描述性统计结果,若 AE 发生率低(如 $\leq 5\%$ )且均为 I - II 级轻度反应,可初步认为冲击波治疗在本研究人群中安全性良好(分别统计 I 、II 、III、IV级 AE 的患者数占总患者数的比例)。

### 六、研究干预\*

6.1 研究干预内容(干预内容的描述、实施步骤、干预药物的剂量与给药途径、 干预的频率频次、试验组和对照组的产品等)

试验组:第1天行第一次髌腱联合筋膜手法协调中心点体外冲击波治疗,1 周后行第二次髌腱联合筋膜手法协调中心点体外冲击波治疗,2周后行第三次髌 腱联合筋膜手法协调中心点体外冲击波治疗。

对照组:第1天行第一次单纯髌腱体外冲击波治疗,1周后行第二次单纯髌腱体外冲击波治疗,2周后行第三次单纯髌腱体外冲击波治疗。

髌腱联合筋膜手法协调中心点体外冲击波干预方法:首先,由筋膜治疗师给患者进行患侧下肢筋膜评估,确定患者患侧下肢有可能导致髌腱炎症状的致密的协调中心点,并用马克笔标记。接下来,由负责冲击波治疗的另一名治疗师给患者进行冲击波治疗。患者仰卧在治疗床,患侧膝关节屈曲 90°固定。在髌腱处进行冲击波治疗(比利时 Gymna Shock Master 500 体外冲击波治疗仪),频率为8Hz,能量为2.0Bar,共2000次。休息1分钟后,在髌腱处进行总共4000次安慰剂冲击波治疗。再休息1分钟后,在筋膜治疗师评估后标记的协调中心点处进行冲击波治疗(比利时 Gymna Shock Master 500 体外冲击波治疗仪),频

率为 8Hz,能量为 2.0Bar,总共 4000 次冲击治疗。患者一共进行 3 次疗程,每次疗程之间间隔 1 周。在治疗前和全部治疗结束后当天对所有受试者进行评估,并于全部治疗结束后第 1 个月和第 3 个月对所有受试者进行随访。

单纯髌腱冲击波干预方法:患者仰卧在治疗床,患侧膝关节屈曲 90°固定。在髌腱处进行冲击波治疗(比利时 Gymna Shock Master 500 体外冲击波治疗仪),频率为 8Hz,能量为 2.0Bar,共 2000 次。休息 1 分钟后,在髌腱处进行总共4000 次同样的冲击波治疗。再休息 1 分钟后,在筋膜治疗师评估后标记的协调中心点处进行总共4000 次安慰剂冲击波治疗。患者一共进行 3 次疗程,每次疗程之间间隔 1 周。在治疗前、全部治疗结束后当天对所有受试者进行评估,并在全部治疗结束后第 1 个月和第 3 个月进行随访。

- 6.2 准备/处理/储存/职责(当干预为药物时,应明确药物与对照品的分配计划) 所需仪器设备均已备齐,均存放于本科,由专门人员负责。
- 6.3 研究干预依从性(如何保持、评价并验证研究的依从性) 充分与患者沟通,使患者能够完成治疗疗程。
- 6.4 合并治疗(被允许的辅助性用药、补充/替代疗法) 冲击波治疗的合并治疗方案<sup>[18]</sup>如下:

第一阶段(1-3周,治疗期):每周一次冲击波治疗合并每日进行单腿(患侧)深蹲的离心康复训练(每日30min,分3次完成)。

第二阶段(4-12 周,随访期)(如第一阶段疼痛下降〈30%):停止冲击波治疗,继续每日进行单腿(患侧)深蹲的离心康复训练(每日 30min,分 3 次完成)。

被允许的补充疗法:在研究期间如患者疼痛明显加重,可允许治疗后 10-15 分钟局部冰敷治疗。

6.4.1 抢救(药物、治疗方式、相关记录.....)

研究期间给予患者干预或评估时, 密切观察情况, 及时处理。

在冲击波治疗过程,如患者出现痛性眩晕、明显冷汗、最低强度仍然难以耐 受疼痛等反应,应立即停止操作,让患者治疗床上仰卧,测量血压、心率、指尖 血糖等,必要时给予保暖、喝糖水以及静脉输液。 七、研究干预中止/受试者中止和退出\*

7.1 研究干预中止(暂时中止的原因/标准:如出现多少不良事件、中止研究的时间长短、在中止研究期间如何收集数据以及如何重新启用研究干预、中止干预期间是否继续随访)

### 中止标准:

- 1. 安全性问题:如果研究过程中出现严重的不良事件、安全性问题或伦理问题,可能危及受试者的健康和安全,或者违反了伦理原则研究应当立即中止或终止。
- 2. 疗效不足:如果研究结果显示治疗措施无效或者疗效不明显甚至对受试者有害,研究者应该考虑中止或终止该研究。
- 3. 研究违反伦理原则:伦理原则是临床研究的基础,如果研究违反了伦理原则,例如未得到受试者知情同意、对受试者隐瞒重要信息等,研究应当立即中止或终止。
- 4. 研究进度缓慢:如果研究进度缓慢,无法按计划完成研究,研究者可考虑中止或终止研究。
- 5. 疾病进展: 若患者病情在治疗期间出现明显恶化, 甚至需要转为外科手术或其他更侵入性治疗, 也应终止冲击波方案。

中止时长:研究中止的持续时间视具体情况而定,通常为2至4周以进行充分的数据评估和专家委员会审查。

数据收集:在中止期间,研究团队仍将通过预定随访计划收集安全性数据和 受试者反馈,以全面了解干预暂停对受试者的潜在影响。所有数据均纳入最终统 计分析。

重新启动标准:在获得伦理委员会的批准和专家组确认安全性评估通过后, 干预措施将在短期内重新启用。研究团队将根据重新启动时的安全性评估结果, 适当调整干预剂量或频率以降低潜在风险。

中止干预期间的随访:在干预暂时期间,研究团队将继续按照原定随访计划 收集受试者的临床数据和主观反馈。随访内容包括但不限于不良事件的记录、疼 痛评分、功能评估和日常活动的监测。

7.2 受试者中止/退出研究(受试者中止试验的可能原因; 涉及植入性器械, 讨

论怎么取出/替代,替代材料的获取,与受试者的后期联系等)

- 1. 患者出现冲击波治疗过程中或治疗后,疼痛反应严重,严重痛性晕厥并且无法再耐受治疗等不良事件;
- 2. 患者中途出现依从性差、主动退出或自行更换其他治疗方案的情况,同样构成终止条件。
- 7.3 失访(减少失访和减少因失访导致数据缺失的措施)
- 1. 临床试验进行过程中,记录治疗期间及治疗随访期间发生的所有自感异常的症状、持续时间、严重度、相应处理措施、转归、对原发病的影响,与治疗的相关性以及对不良反应的整体评价;
- 2. 提前跟患者讲明试验要求,并签署知情同意书,为了确保高随访率,负责人员需要登记各入选患者及两个或以上的亲属的联系方式,包括姓名、电话(移动电话和固定电话)、联系地址、电子邮箱。按照各随访时间点定期要求患者需前往门诊进行随访。

### 八、不良事件和非预期事件

- 8.1 不良事件
- 8.1.1 不良事件的定义(必须详细写出不良事件涉及的各项指标)
  - 1. 治疗过程中不良事件

冲击波治疗过程中局部疼痛或不适, 甚至出现心率加快、冷汗、痛性晕厥等。

- 2. 治疗后不良事件
- (1) 冲击波治疗后局部短暂疼痛加重等;
- (2) 冲击波治疗后局部淤血、轻度肿胀等;
- (3)冲击波治疗后局部皮肤红斑。

### 8.1.2 不良事件的分类

分为治疗过程中、治疗后不良事件,治疗操作相关及个体差异相关不良事件。 8.1.3 不良事件的评价(不良事件的严重程度、不良事件与研究的相关性、不良事件是否为研究干预已知的不良事件等)

根据受试者的临床症状评估是否出现不良事件以及不良事件的严重程度,判断是治疗相关或是个体差异相关的不良事件。

### 8.1.4 不良事件的报告

发生不良事件 24 小时内及时上报研究项目负责人,根据不良事件的严重程 度按照孙逸仙纪念医院的相关规定上报相关部门。

- 8.2 严重不良事件
- 8.2.1严重不良事件的定义
  - 1. 治疗过程中严重不良事件

冲击波治疗过程中疼痛反应极其明显,甚至出现心率明显加快、休克、晕厥等,且停止治疗后症状并未逐渐减轻。

- 2. 治疗后严重不良事件
- (1) 冲击波治疗后皮肤破溃, 甚至出现感染等;
- (2) 冲击波治疗后深层组织损伤、血管破裂等;
- (3) 冲击波治疗后神经损伤等。

### 8.2.2 严重不良事件的分类

分为治疗过程中、治疗后严重不良事件,治疗操作相关及个体差异相关严重 不良事件。

### 8.2.3 严重不良事件的评价

根据受试者的临床症状评估是否出现严重不良事件,判断是治疗相关或是个体差异相关的严重不良事件。

#### 8.2.4 严重不良事件的报告

发生严重不良事件 24 小时内及时上报研究项目负责人并按照孙逸仙纪念医院的相关规定 24 小时内报告伦理委员会,并按照研究方案的规定随访,及时提交随访报告。

- 8.3 特殊权益事件
- 8.3.1 特殊权益事件的定义

冲击波治疗研究本身相关的具有特定科学和医学关注价值的事件。

#### 8.3.2 特殊权益事件的分类

分为特殊人群(如老年人)相关特殊权益事件、心血管事件相关特殊权益事件和治疗部位反应(如局部组织反应明显)相关特殊权益事件。

### 8.3.3 特殊权益事件的评价

根据受试者的个体差异和临床症状评估是否出现特殊权益事件事件,判断是治疗相关或是个体差异相关的特殊权益事件。

### 8.3.4 特殊权益事件的报告

发生特殊权益事件 24 小时内及时上报研究项目负责人,持续监测并根据严重程度看是否需要按照孙逸仙纪念医院的相关规定 24 小时内报告伦理委员会,并按照研究方案的规定随访,及时提交随访报告。

### 8.4 非预期事件

#### 8.4.1 非预期事件的定义

冲击波治疗研究期间出现的、未在研究方案的已知不良事件清单中列明,且 与冲击波治疗的潜在风险相关的任何不良医学事件,比如头痛等。

### 8.4.2 非预期事件的分类

分为非严重非预期事件和严重非预期事件。

### 8.4.3 非预期事件的评价

根据患者的临床症状评估是否出现非预期事件事件,判断是治疗时间、强度 可能相关或是个体差异(生理)可能相关的非预期事件。

#### 8.4.4 非预期事件的报告

发生严重非预期事件 24 小时内及时上报研究项目负责人并按照孙逸仙纪念 医院的相关规定 24 小时内报告伦理委员会,并按照研究方案的规定随访,及时 提交随访报告。发生非严重非预期事件 24 小时内及时上报研究项目负责人并根 据受试者具体情况进行处理。

### 九、数据收集及管理

### 9.1 病例报告表/电子数据记录

采用中山大学孙逸仙纪念医院临床研究病例报告表详细记录受试者的研究编号和基本信息、临床研究的流程图、入选标准、排除标准、受试者的既往病史、基线的相关检查和指标评估、治疗后的相关检查和指标评估、随访1个月和随访3个月的相关检查和指标评估、合并用药表、不良事件记录表、严重不良事件记录表和研究完成情况的总结。

9.2 数据管理(数据的采集形式、数据存储载体:电子/纸质、数据完整性检验、数据库建立方法、数据管理系统、数据质量检测方法、数据锁库的定义等)

依据中山大学孙逸仙纪念医院临床研究病例报告表,使用 RedCap 制定电子病例报告表,并在系统中配置字段、数据类型、必填规则和范围检查。在投入使用前进行功能验证,并对相关统计人员进行基于角色的系统与电子病例报告表培训,确保每位用户仅能访问其职责范围内的数据。收集纸质数据(源数据)后,现场工作人员通过安全的 Web 界面实时输入源数据(源文件 → eCRF),系统自动执行实时编辑检查。对关键变量采用双人独立录入或抽样复核,以降低键入错误率。所有数据在传输过程中采用 TLS 加密,存储在符合 GCP 与 FDA 21 CFR Part 11 要求的受控服务器上,并定期进行备份与灾备演练。

提高数据质量的方法:

系统内置范围、逻辑、一致性等自动校验规则,录入时即时提示错误,录入 后生成查询供监测人员处理;

每一次数据创建、修改、删除均记录用户、时间、操作类型,满足监管审计需求:

监查员对关键变量进行现场或远程核对,确保电子记录与原始数据一致;

数据管理团队定期导出数据进行统计检查(缺失、异常分布),并通过查询/答复循环解决不一致:

依据关键风险指标(关键变量缺失率、编辑检查触发率)动态调整监查频次, 提高效率。

在所有查询解决、数据清理完成后,依据 SOP 进行正式锁定,锁定后任何 更改必须经批准并记录在案。

整个过程需编制并维护《系统验证报告》《数据管理手册》《编辑检查手册》等文档,以备监管审查。

### 十、伦理学要求

本研究遵守《药物临床试验质量管理规范》 以及 《医疗卫生机构开展研究者发起的临床研究管理办法》(试行)的规定及赫尔辛基宣言。试验开始之前,由我院伦理委员会的批准该方案后方可开展本项研究。在研究过程中,如果必须进行方案修订,修订后方案必须重新递交伦理委员会审查,研究者必须等到伦理委员会同意意见后方可执行新方案。

每个入组病人必须签署知情同意书。知情同意书的复印件和研究者及伦理委员会的联系方式必须提供给受试者\*。本研究会收集研究对象的临床资料、个人信息用以进行科学研究,会涉及患者的隐私权益。本研究参加人员及数据分析人员均签署保密合同,不向任何与本研究无关的个人和机构泄露患者个人信息及疾病相关信息。所收集的患者数据实施统一管理,杜绝个人隐私外泄。

### 十一、参考文献

- [1] Rudavsky A, Cook JL, Docking S (2018) .Proximal patellar tendon pathology can develop during adolescence in young ballet dancers—a 2 year longitudinal study. Scand J Med Sci Sports 28:2035–2041.
- [2] Peers KH, Lysens RJ (2005) Patellar tendinopathy in athletes:current diagnostic and therapeutic recommendations. Sport Med 35:71–87.
- [3] Larsson ME, Kall I, Nilsson-Helander K. Treatment of patellar tendinopathy—a systematic review of randomized controlled trials[J]. Knee Surg Sports Traumatol Arthrosc, 2011, 20(8): 1632-1646.
- [4] Qassim I Muaidi .Rehabilitation of patellar tendinopathy.J Musculoskelet Neuronal Interact. 2020 Dec 1;20(4):535-540.
- [5] Furia JP, Rompe JD, Cacchio A, et al. A single application of low-energy radial extracorporeal shock wave therapy is effective for the management of chronic patellar tendinopathy[J]. Knee Surg Sports Traumatol Arthrosc, 2013, 21(2): 346-350.
- [6] Zwerver, J., & Dekker, F. . Patient guided Piezoelectric Extracorporeal Shockwave Therapy as treatment for chronic severe patellar tendinopathy: A pilot study. Journal of Back and Musculoskeletal Rehabilitation, 2010, 23(3), 111–113.
- [7] Peers, K. H. . Extracorporeal shock wave therapy in chronic patellar tendinopathy: a randomised double-blinded, placebo-controlled trial. British Columbia Medical Journal, 2003, 45(9), 500–505.
- [8] Yan, H. M., & Meng, Q. S.. Observation on the efficacy of extracorporeal shock wave therapy for patellar tendinitis in 48 cases. Zhejiang Traumatic Surgery, 2019, 24(4), 730–737.
- [9] Geng, J. B., Li, M. Q., & Peng, Q. J. . Clinical evaluation of small needle knife combined with extracorporeal shock wave for patellar tendinitis. World Journal of Traditional Chinese Medicine, 2017, 12(9), 2172–2173.
- [10]中国研究型医院学会冲击波医学专业委员会. 中国骨肌疾病体外冲击波疗法指南(2023 年版) [J].中国医学前沿杂志(电子版), 2023, 15(9): 1-10.
- [11]中华医学会物理医学与康复学分会,肌肉骨骼疾病体外冲击波治疗专家共识组.肌肉骨骼疾 病体外冲击波治疗专家共识[J].中华物理医学与康复杂志,2019,41(7):481-487.
- [12] van Leeuwen MT, Zwerver J, van den Akker-Scheek I. Extracorporeal shockwave therapy for patellar tendinopathy: a review of the literature[J]. Br J Sports Med, 2009, 43(3): 163-168.

- [13] Rhim HC, Shin J, Kang J, et al. Use of extracorporeal shockwave therapies for athletes and physically active individuals: a systematic review. Br J Sports Med 2024;58:154–63.
- [14] Schroeder AN, Tenforde AS, Jelsing EJ. Extracorporeal Shockwave Therapy in the Management of Sports Medicine Injuries. Curr Sports Med Rep 2021;20:298–305.
- [15] Liu, L., Huang, Q. M., Liu, Q. G., et al. . Research progress on myofascial trigger point theory and its application in sports rehabilitation. Chinese Journal of Rehabilitation Theory and Practice, 2016, 22(10), 1167–1170.
- [16] Alessandro Pedrelli, Carla Stecco, Julie Ann Day. Treating patellar tendinopathy with Fascial Manipulation. J Bodyw Mov Ther. 2009 Jan;13(1):73-80.
- [17] Johannes Zwerver, Evert Verhagen, Fred Hartgens, Inge van den Akker-Scheek, Ron L Diercks. The TOPGAME-study: effectiveness of extracorporeal shockwave therapy in jumping athletes with patellar tendinopathy. Design of a randomised controlled trial. BMC Musculoskelet Disord. 2010 Feb 8:11:28.
- [18] DRAGOO J L, WASTERLAIN A S, BRAUN H J, et al. Platelet- rich plasma as a treatment for patellar tendinopathy: a double-blind, randomized controlled trial [J]. Am J Sport Med, 2014, 42 (3): 610-618.

### 1. 流程图示例



## 2. 研究日程表示例

| 程序 | 筛选期-7<br>至-1 天 | 入组/基<br>线访视 1<br>第 1 天 | 入组/基<br>线访视 2<br>第 8±1<br>天 | 入组/基<br>线访视 3<br>第 15±1<br>天 | 入组/基<br>线访视 4<br>第 45±1<br>天 | 入组/基<br>线访视 5<br>第 75±1<br>天 | 研究结束<br>访视 6<br>第 105±<br>1 天 |
|---|---|---|---|---|---|---|---|
| 知情同意<br>书 | √ | | | | | | |
| 人口统计 学 | <b>√</b> | | | | | | |
| 病史 | √ | | | | | | |
| 体格检查 | √ | | | | | | |
| 伴随用药<br>史回顾 | V | | | | | | |
| 影像学检查 | V | | | | | | |
| 随机 | √ | | | | | | |
| 研究干预 | | √ | √ | √ | | | |
| VAS 评分 | √ | | | √ | √ | | √ |
| Lysholm<br>膝关节<br>评分 | V | | | <b>V</b> | V | | √ |
| 髌腱厚度 | √ | | | √ | | | |
| 不良事件<br>回顾与评<br>估 | V | <b>V</b> | <b>V</b> | <b>√</b> | <b>V</b> | <b>V</b> | √ |
| 完成病例 报告表 | V | V | V | V | V | V | V |